CLINICAL TRIAL: NCT04336059
Title: Pericapsular Nerve Group Block in Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: hip arthroplasty
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2020-12

CONDITIONS: Post Operative Pain After Hip Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Other): will receive sham PENG block with normal saline in total volume of 20 ml.
  Interventions: Procedure: pericapsular nerve group block
- group 2 (Experimental): will receive real PENG block with bupivacaine (0.25%) in total volume of 20 ml.
  Interventions: Procedure: pericapsular nerve group block

INTERVENTIONS:
Procedure: pericapsular nerve group block — The regional block will be performed with the patient in the supine position under complete sterile technique. A low frequency curvilinear ultrasound probe will be initially placed in a transverse plane over the anterior inferior iliacspine (AIIS) and then aligned with the pubic ramus by rotating the probe counterclockwise approximately 45 degrees. In this view, the iliopubic eminance(IPE), the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle will observed.
  A 22-gauge, 80-mm needle will be inserted from lateral to medial in an in-plane approach to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly after local infiltration of the site of the block with 3 ml lidocaine 2%. Following negative aspiration,the normal saline solution will injected in 5-mL increments while observing for adequate fluid spread in this plane.

SUMMARY:
Peripheral nerve blocks are becoming increasingly popular for hip surgery anesthesia. Modern regional anesthesia for major hip surgery includes the use of a single shot and continuous epidural or spinal injections, continuous lumbar plexus blockade and continuous peripheral blockade of the femoral nerve (FN), fascia iliaca (FI) block, 3-in-1 FN block and sciatic nerve. The use of either single shot or continuous peripheral nerve blocks are becoming increasingly popular.

This study will be conducted to evaluate the effect of ultrasound guided pericapsular nerve group block in hip arthroplasty surgery.

DETAILED DESCRIPTION:
Hip joint is richly innervated, and the pain following hip arthroplasty is particularly severe. Effective postoperative analgesic technique especially in an elderly with significant comorbidities is challenging. (1) Peripheral nerve blocks are becoming increasingly popular for hip surgery anesthesia. Modern regional anesthesia for major hip surgery includes the use of a single shot and continuous epidural or spinal injections, continuous lumbar plexus blockade and continuous peripheral blockade of the femoral nerve (FN), fascia iliaca (FI) block, 3-in-1 FN block and sciatic nerve. The use of either single shot or continuous peripheral nerve blocks are becoming increasingly popular. (2) These techniques have shown effective and safe postoperative pain control, resulting in lower opioid consumption, improved earlier rehabilitation and high patient satisfaction. (3) Pericapsular nerve group (PENG) block has been recently recommended by Giron-Arango et al. for use as postoperative analgesia in hip surgeries. It is a new regional anesthesia method based on blocking the articular branches of femoral nerve (FN) and accessory obturator nerve(AON) and obturator nerve in the region between the anterior inferior iliac spine (AIIS) and ilio-pubic eminence (IPE).The anterior capsule is the most richly innervated section of the joint suggesting these nerves should be the main targets for hip analgesia. (4)

ELIGIBILITY:
Inclusion Criteria:

* Patients will involve in the research if they will schedule for unilateral hip arthroplasty (THA) surgery.
* aged more than 50 years of both genders.
* have American society of anesthiologists physical status I-II and III.

Exclusion Criteria:

* Revision hip arthroplasty.
* hip arthroplasty. combined with subtrochanteric shortening osteotomy.
* drug allergy.
* regular narcotic use.
* renal &/ or hepatic impairments.
* coagulopathy disorders.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
first time of rescue analgesia. | postoperative first day
  first time of rescue morphine analgesia.

SECONDARY OUTCOMES:
postoperative morphine consumption | postoperative first day
  postoperative morphine consumption as rescue analgesia
pain score | postoperative first day
  pain score by numerical rating score

CONTACTS AND LOCATIONS:
Locations (1):
- Tarek Abdel Hay, Tanta, El Gharbyia, Egypt

IPD SHARING:
Plan to Share IPD: No